CLINICAL TRIAL: NCT06708806
Title: Cell Ongrowth and Biocompatibility Study of Two Different (Hydrophobic Acrylic) Intraocular Lenses: IOL XY1 vs. IOL XY1A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Leydolt, Assoc. Prof. Priv. Doz. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HOPP; 2060/2019 (Other: Medical University of Vienna - Ethic Committee)
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cataract
Keywords: Biocompatibility
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of the biocompatibility of two different IOLs. Investigated IOLs will be implanted subsequently according to the study protocol with one IOL type in the eye with no astigmatism and the other IOL type in the eye with astigmatism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toric vs Monofocal IOL (Other): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm one (I) participants will receive a monofocal IOL (XY1) vs. an toric IOL (XY1A)
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (XY1) vs. an toric IOL (XY1A)

SUMMARY:
The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral randomized IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved investigational plan.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation is planned
* Age 40 and older
* Astigmatism of at least 0.75Diopters in one eye
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Diabetes mellitus
* Pseudoexfoliation syndrome
* Systemical anticoagulation
* Antiphlogistic therapy
* Antiglaucomatosa
* Uncontrolled systemic or ocular disease
* Preceding ocular surgery or trauma
* Intraoperative complications
* Pregnancy/Nursing
* Concurrently participating in any other clinical trial or if they have participated in any other clinical trial during the last 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Foreign Body Giant Cells | 6 weeks
  The primary objective is to assess the difference in Foreign Body Giant Cells between monofocal and toric lenses in every patient at 6 weeks follow up.

SECONDARY OUTCOMES:
Foreign Body Giant Cells | 5 months
  The first secondary objective is to assess the difference in Foreign Body Giant Cells between monofocal and toric lenses in every patient at 1 week and 5 months follow up.
small round cells | 5 months
  The second secondary objective is to assess the difference in small round cells between monofocal and toric lenses in every patient at 1 week, 6 weeks and 5 months follow up.
PCO | 5 months
  The third secondary objective is to assess the difference in PCO between monofocal and toric lenses in every patient at 1 week, 6 weeks and 5 months follow up.
anterior chamber reaction | 5 months
  The fourth secondary objective is to assess the difference in the anterior chamber reaction between monofocal and toric lenses in every patient at 1 week, 6 weeks and 5 months follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided